CLINICAL TRIAL: NCT06231160
Title: Clinical Comparative Study of Systematic Therapy Combined With Microwave Ablation and Systematic Therapy for Pancreatic Cancer
Brief Title: Clinical Comparative Study of Systematic Therapy Combined With MWA and Systematic Therapy for Pancreatic Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Ping Liang, Director, Chinese PLA General Hospital
Other Study IDs: 82171941
Record Dates: First submitted 2023-12-24; First posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Pancreatic Neoplasms; Ablation
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Systematic Therapy Combined With Microwave Ablation: Perform microwave ablation for patients with pancreatic cancer, and then conduct chemotherapy according to the guidelines two to three weeks later
  Interventions: Procedure: Systematic Therapy Combined With Microwave Ablation
- Systematic Therapy: Using the same chemotherapy method as the experimental group

INTERVENTIONS:
Procedure: Systematic Therapy Combined With Microwave Ablation — Patients with unresectable pancreatic cancer were included for laboratory examination, and quality of life and pain scores were recorded. The experimental group underwent microwave ablation first, followed by chemotherapy according to the guidelines; The control group received the same chemotherapy. Record the use of chemotherapy drugs and the occurrence of adverse events. Follow up will be conducted at 30 days, 90 days, and 180 days after chemotherapy to evaluate pancreatic function and quality of life.
  Other Names: Systematic Therapy
  Groups: Systematic Therapy Combined With Microwave Ablation

SUMMARY:
Pancreatic carcinoma (PC) is the deadliest malignant tumors worldwide. Surgical resection is one of the most effective methods for the treatment of PC, but the resectable rate is less than 20% among the patients with PCs, and the recurrent and metastatic rate is more than 80% in two years after resection. Ablation has been confirmed one of the most effective methods for solid tumors by recent twenty years and proven to be a radical treatment similar to the surgical resection for the clinical applications of hepatic and renal tumors at early clinical staging in the internationally guidelines. The purpose is to explore the efficacy and safety of microwave ablation in the treatment of pancreatic cancer in combination with systematic therapy.

DETAILED DESCRIPTION:
Pancreatic carcinoma (PC) is the deadliest malignant tumors worldwide. Surgical resection is one of the most effective methods for the treatment of PC, but the resectable rate is less than 20% among the patients with PCs, and the recurrent and metastatic rate is more than 80% in two years after resection. Furthermore, it is difficult to achieve tumoral complete responses by traditional therapies including chemotherapy, radiotherapy and transarterial embolization. Ablation has been confirmed one of the most effective methods for solid tumors by recent twenty years and proven to be a radical treatment similar to the surgical resection for the clinical applications of hepatic and renal tumors at early clinical staging in the internationally guidelines. However, the published clinical practices on the thermal ablation of PCs with large-scale cases are rare. One of the most important reasons for this originates from the extreme complexity and difficult regulation of the temperature distribution in tumors during thermal ablation because of the own characteristics of PCs, including highly invasive growth without tumoral capsules, high proportion of the interstitial fiber tissue, and the unusual blood perfusion because of extremely chaotic microvascular structures. The purpose is to explore the efficacy and safety of microwave ablation in the treatment of pancreatic cancer in combination with systematic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Inoperable pancreatic cancer
* Age from 18 to 80
* PS score from 0 to 3
* Clear pathological diagnosis

Exclusion Criteria:

* Severe coagulation dysfunction
* Individuals with severe heart, lung, liver, and kidney dysfunction
* Individuals with acute or active infectious lesions in any part of the body
* Researchers believe that there are any other factors that are not suitable for inclusion or that affect the participation of participants in the study
* Psychological health issues that hinder this experiment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pancreatic cancer
Sampling Method: Non-Probability Sample
Enrollment: 185 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
overall survival | 30, 90, and 180 days after the end of the last chemotherapy
  Time from receiving treatment to death

SECONDARY OUTCOMES:
Pain relief rate | 30, 90, and 180 days after the end of the last chemotherapy
  Pain relief before and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ping Liang, Study Chair — The Fifth Medical Center of the General Hospital of the PLA of China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Siegel RL, Miller KD, Wagle NS, Jemal A. Cancer statistics, 2023. CA Cancer J Clin. 2023 Jan;73(1):17-48. doi: 10.3322/caac.21763. PMID 36633525
- [Background] Kluger MD, Epelboym I, Schrope BA, Mahendraraj K, Hecht EM, Susman J, Weintraub JL, Chabot JA. Single-Institution Experience with Irreversible Electroporation for T4 Pancreatic Cancer: First 50 Patients. Ann Surg Oncol. 2016 May;23(5):1736-43. doi: 10.1245/s10434-015-5034-x. Epub 2015 Dec 29. PMID 26714959
- [Background] Wang Z, Liu M, Zhang DZ, Wu SS, Hong ZX, He GB, Yang H, Xiang BD, Li X, Jiang TA, Li K, Tang Z, Huang F, Lu M, Chen JA, Lin YC, Lu X, Wu YQ, Zhang XW, Zhang YF, Cheng C, Ye HL, Wang LT, Zhong HG, Zhong JH, Wang L, Chen M, Liang FF, Chen Y, Xu YS, Yu XL, Cheng ZG, Liu FY, Han ZY, Tang WZ, Yu J, Liang P. Microwave ablation versus laparoscopic resection as first-line therapy for solitary 3-5-cm HCC. Hepatology. 2022 Jul;76(1):66-77. doi: 10.1002/hep.32323. Epub 2022 Jan 28. PMID 35007334
- [Background] Fegrachi S, Walma MS, de Vries JJJ, van Santvoort HC, Besselink MG, von Asmuth EG, van Leeuwen MS, Borel Rinkes IH, Bruijnen RC, de Hingh IH, Klaase JM, Molenaar IQ, van Hillegersberg R. Safety of radiofrequency ablation in patients with locally advanced, unresectable pancreatic cancer: A phase II study. Eur J Surg Oncol. 2019 Nov;45(11):2166-2172. doi: 10.1016/j.ejso.2019.06.008. Epub 2019 Jun 12. PMID 31227340
- [Background] Martin RC 2nd, Kwon D, Chalikonda S, Sellers M, Kotz E, Scoggins C, McMasters KM, Watkins K. Treatment of 200 locally advanced (stage III) pancreatic adenocarcinoma patients with irreversible electroporation: safety and efficacy. Ann Surg. 2015 Sep;262(3):486-94; discussion 492-4. doi: 10.1097/SLA.0000000000001441. PMID 26258317
- [Background] Vogl TJ, Panahi B, Albrecht MH, Naguib NNN, Nour-Eldin NA, Gruber-Rouh T, Thompson ZM, Basten LM. Microwave ablation of pancreatic tumors. Minim Invasive Ther Allied Technol. 2018 Feb;27(1):33-40. doi: 10.1080/13645706.2017.1420664. Epub 2017 Dec 26. PMID 29278340